CLINICAL TRIAL: NCT07001644
Title: Microneedling Versus Carboxytherapy Either With or Without Platelet Rich Plasma in Treating Stria Distensae Rubra
Brief Title: Microneedling Versus Carboxytherapy in Stria Distensae Rubra
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0107162
Record Dates: First submitted 2025-05-17; First posted 2025-06-03 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2024-10

CONDITIONS: Striae Distensae
Keywords: striae distensae; striae rubra; microneedling; carboxytherapy
MeSH Terms: conditions — Striae Distensae | interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treated with microneedling (Active Comparator): microneedling with topical application of PRP on one side of abdomen and microneedling only on the other side
  Interventions: Device: microneedling
- treated with carboxytherapy (Active Comparator): carboxytherapy with intradermal injection of PRP on one side of abdomen and carboxytherapy only on the other side
  Interventions: Device: Carboxytherapy

INTERVENTIONS:
Device: microneedling — microneedling with topical application of PRP on one side of abdomen and microneedling only on the other side.
  Arms: treated with microneedling
Device: Carboxytherapy — carboxytherapy with intradermal injection of PRP on one side of abdomen and carboxytherapy only on the other side.
  Arms: treated with carboxytherapy

SUMMARY:
The aim of this study is to evaluate and compare the efficacy and safety of microneedling and carboxytherapy either with or without platelet-rich plasma in the treatment of striae distensae rubra.

ELIGIBILITY:
Inclusion Criteria:

* Female patients.
* Age ranging from 18-45 years old.
* Fitzpatrick skin type III-IV.
* Striae distensae rubra on the abdomen (bilateral and more or less symmetrical).

Exclusion Criteria:

* Patients taking immunosuppressants or having any disease affecting wound healing including diabetes.
* Patients receiving systemic glucocorticoids for chronic health conditions.
* Patients with chronic dermatologic diseases such as psoriasis and vitiligo.
* Pregnant and lactating females.
* Patients with a tendency for keloid formation.
* Patients with endocrine disturbance.
* Patients with autoimmune diseases, systemic diseases such as severe anemia, respiratory, cardiac, renal or liver disorder.
* Patients with bleeding and coagulation disorders.
* Patients who received any form of treatment for their SD in the past 6 months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in the size of the stria distensae rubra | group I: six sessions over 18 weeks , group II: 6 sessions over 12 weeks, followed in both groups by three months of follow up
  will be assessed by digital photography, actual measurement of the stria before and after treatment, and objective assessment of the percent of improvement

CONTACTS AND LOCATIONS:
Overall Officials: professor doctor Amira Eid, Principal Investigator — Alexandria University
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided